CLINICAL TRIAL: NCT07365488
Title: Effect of Virtual Reality Versus Binaural Beat Stimulation on Sleep Disturbances and Patient Discomfort Following Prosthetic Mechanical Valve Replacement Surgery: A Randomized Controlled Trial
Brief Title: Effect of Virtual Reality and Binaural Beat on Sleep and Comfort in Adults After Mechanical Valve Replacement Surgery
Acronym: VR-BBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahraa Qasem Karem (Other)
Responsible Party: Sponsor-Investigator, Zahraa Qasem Karem, Zahraa Qasem, MSc Nursing, University of Baghdad, Adult Nursing, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VRBBS-MVR-SOUND-OF-THE- VALVE; 24-18-Nov-2025 (Other: University of Baghdad , College of Nursing Research Ethics Committee)
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Patients Following Prosthetic Mechanical Valve Replacement, Focusing on Sleep Disturbances and Patient Discomfort
Keywords: Prosthetic Mechanical Valve Replacement , Mechanical valve sound , Sleep Dist

STUDY DESIGN:
Intervention Model Description: 1. VR Group - receiving a Virtual Reality relaxation sessiones.
  2. Binaural Beat Group - receiving a Binaural Beat Stimulation sessions.
  3. VR + Binaural Beat Group - receiving both interventions.
  4. Control Group - receiving standard postoperative care without interventionsز
  Randomization ensures that each participant has an equal chance of being assigned to any group, and all groups are followed concurrently to compare outcome.
Masking Description: Not applicable - study is open label; all participants and staff are aware of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VR Group (Experimental): Guided VR relaxation sessions
  Interventions: Behavioral: Virtual Reality Relaxation
- Binaural Beat Group (Experimental): sessions BBS for reducing discomfort and enhance sleep quality
  Interventions: Behavioral: Binaural Beat Stimulation
- VR + Binaural Beat Group (Experimental): Combined VR & BBS sessions
  Interventions: Behavioral: VR + Binaural Beat Group
- Control Group (Other): Standard postoperative care
  Interventions: Other: Standard Postoperative care

INTERVENTIONS:
Behavioral: Virtual Reality Relaxation — Guided VR relaxation sessions to reduce discomfort an enhance sleep quality
  Arms: VR Group
Behavioral: Binaural Beat Stimulation — Guide sessions BBS to reduce discomfort and enhance sleep quality
  Arms: Binaural Beat Group
Behavioral: VR + Binaural Beat Group — Combined VR & BBS sessions
  Arms: VR + Binaural Beat Group
Other: Standard Postoperative care — Usual postoperative care for patients
  Arms: Control Group

SUMMARY:
This study will compare the effects of Virtual Reality and Binaural Beat Stimulation on sleep quality and discomfort in adult patients who have undergone prosthetic mechanical valve replacement surgery. Many patients experience sleep disturbances and discomfort due to the sound of the mechanical valve. Participants will be randomly assigned to one of two non-drug interventions to see which method improves sleep and reduces discomfort after surgery. The study aims to help improve recovery and comfort for patients after valve replacement.

DETAILED DESCRIPTION:
This randomized clinical trial will evaluate the effects of four interventions on sleep disturbances and patient discomfort in adult patients after prosthetic mechanical valve replacement. Sleep disturbances are common due to the sound of the mechanical valve. Participants will be randomly assigned to one of four groups: (1) VR Group (2) Binaural Beat Group listening to binaural beats for 20 minutes (3) VR + Binaural Beat Group combining both interventions, and (4) Control Group receiving standard postoperative care without interventions. Primary outcomes include sleep quality and patient-reported discomfort measured during the early postoperative period. The study aims to identify which intervention or combination is most effective in improving recovery and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for participation following mechanical valve replacement surgery if they are willing to participate, able to provide informed consent, and meet the following criteria: male or female aged 18 years or older, hemodynamically stable, oriented and conscious without cognitive impairment, free from visual or auditory impairments, able to communicate orally in Arabic, not receiving analgesics or sedatives within at least four hours prior to the intervention, and having no history of epilepsy, seizure disorders, or recurrent migraines.

Exclusion Criteria:

* The study's exclusion criteria will include participants with facial or head injuries, a history of vertigo or severe motion sickness, immediate postoperative cardiac arrest, the use of hypnotic medications, the presence of a tracheostomy, or any implanted body hardware.

Ages: 28 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Patient Discomfort | From postoperative day 3 until discharge from the cardiac surgery ward
  Patient-reported discomfort measured using the Kolcaba Verbal Rating Comfort Scale (KCS), assessing the intensity of postoperative discomfort following prosthetic mechanical valve replacement. This measure captures the level of discomfort experienced by the patient during hospitalization that result from mechanical valve sound.

CONTACTS AND LOCATIONS:
Overall Officials: Waffa AR Hattab, Ph.D., Principal Investigator — University of Baghdad, College of Nursing
Locations (1):
- Ibn Al-Nafees Teaching Hospital, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Baghdad, College of Nursing — https://www.uobaghdad.edu.iq/
- Available data/document: Study not yet published / Data not available: Study not yet published / Data — https://www.uobaghdad.edu.iq — Study not yet published